CLINICAL TRIAL: NCT03773887
Title: Comparison of Inflammatory Profiles and Regenerative Potential in Alcoholic Liver Disease
Acronym: TargetOH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2014_30; 2014-A01452-45 (Other: ID-RCB Number, ANSM)
Record Dates: First submitted 2018-10-16; First posted 2018-12-12 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Liver Diseases; Acute on Chronic Hepatic Failure
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- acute alcoholic hepatitis (Other): collection of liver biopsies collection of blood samples in patients with acute alcoholic hepatitis (group A)
  Interventions: Other: collection of liver biopsies collection of blood samples
- Alcoholic cirrhosis (Other): collection of liver biopsies collection of blood samples in patients with alcoholic cirrhosis (group B1)
  Interventions: Other: collection of liver biopsies collection of blood samples
- Without chronic liver disease (Other): collection of liver biopsies collection of blood samples in patients without chronic liver disease (group B2)
  Interventions: Other: collection of liver biopsies collection of blood samples

INTERVENTIONS:
Other: collection of liver biopsies collection of blood samples — blood and ascites samples; extraction of explants, hepatic resection parts; hepatic parenchyma on liver biopsies

SUMMARY:
The main objective of this study is the comparison of the profile of the pro-inflammatory cytokines at the patients suffering from an alcoholic hepatitis to that of two groups witnesses: patients suffering from an alcoholic cirrhosis and unhurt patients of chronic liver disease

ELIGIBILITY:
Inclusion Criteria:

* group A: patients with acute alcoholic hepatitis
* Active alcohol abuse defined by DSM IV and excessive alcohol consumption prior to admission (> 60 g per day for men and> 40 g per day for women)
* Moderate elevation of transaminases (less than 500 U / L) with a typical ASAT / ALAT ratio of 2: 1
* Bilirubin> 50 mg / l
* Absence of autoimmune liver disease (ANA <1/80, AML <1/80, LKM1 neg, AAM neg)
* Absence of hepatitis B and C and HIV infection (negative anti-HIV antibodies, negative HBsAg, negative HCV PCR)
* Patients with other acute complications than alcoholic hepatitis may be included (eg, digestive hemorrhage, acute renal failure, infection, etc.)
* Because there is no validated noninvasive tool for the diagnosis of alcoholic hepatitis, histological confirmation is required in all patients (preferably by transjugular biopsy): alcoholic hepatitis will be diagnosed on the presence of the following histological characteristics: Hepatocellular lesions (ballooning, Mallory body)/ Inflammatory infiltrate with polymorphonuclear neutrophils
* group B1: patients with alcoholic cirrhosis
* Decompensated or non-decompensated alcoholic cirrhosis, defined according to the HAS guidelines, ie by a liver biopsy or a cluster of clinico-biological arguments (www.has-sante.fr)
* group B2: patients free from chronic liver disease
* Justification of blood and liver sampling for the management of a pathology other than chronic liver disease (eg liver metastasis of digestive cancer occurring on healthy liver)

Exclusion Criteria:

* For groups A and B1:
* Patients with hepatocellular carcinoma of progressive non-hepatic cancer
* Presence of HBsAg
* Presence of anti-HCV antibodies by positive PCR
* Presence of antibodies to HIV 1 +2
* Pregnancy
* for group B2:
* Alcoholic liver disease
* Presence of HBsAg
* Presence of anti-HCV antibodies by positive PCR
* Presence of antibodies to HIV 1 +2
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
the expression of proinflammatory cytokines | Baseline
  Proinflammatory Cytokines (TNF, IL-1, IL-6, IL-8)

SECONDARY OUTCOMES:
the expression of genetic variants of pro-inflammatory cytokines | Baseline
  Identification of genetic variants of pro-inflammatory cytokines that contribute to mortality of Alcoholic Liver Disease
Cell lysis (AST, ALT, CK18 cleaved) | Baseline
Regeneration markers (Ki-67, Fn14, CK7) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Philppe Mathurin, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez, CHRU, Lille, France